CLINICAL TRIAL: NCT06405620
Title: Mixed Observational Study Evaluating the Use of a Social Assistance Robot in a Population of Children Subjected to Prolonged Isolation
Brief Title: Use of a Social Assistance Robot in a Population of Children Subjected to Prolonged Isolation
Acronym: BUDDY-GUARD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RC31/23/0168
Record Dates: First submitted 2024-04-29; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Social Isolation
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robot intervention (Experimental): the child uses the assistance robot
  Interventions: Other: Assistance robot

INTERVENTIONS:
Other: Assistance robot — the child controls the robot at his parent's home from his room

SUMMARY:
During the period of isolation of the hospitalized child, contacts between the child and his family are impaired. Being away from home as well as from the social and family circle can be harmful for the hospitalized child. It seems necessary to measure the impact of the use of such an assistance robot both on the user himself and his family. Thus, it seems relevant to scientifically validate the benefit of using such an assistance robot to break iatrogenic social isolation and to measure the impact of this use.

ELIGIBILITY:
Inclusion Criteria:

* Children hospitalized in the pediatric hemato-oncology department whose duration of isolation is estimated to be greater than two weeks.
* Children who have accepted the robot and whose parents have accepted its use in their home.
* Agreement of holders of parental authority for the inclusion of the hospitalized child.

Exclusion Criteria:

* Patient or two parents who do not have a sufficient level of French for research.
* Cognitive or motor disorders in children, not allowing the use of the robot and/or the carrying out of semi-structured interviews.
* Cognitive disorders in parents and/or siblings that do not allow semi-structured interviews to be carried out.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the use of a social assistance robot with children hospitalized in the hemato-oncology department and subjected to prolonged isolation | 1 month
  number of activations of the robot and duration of the activations

SECONDARY OUTCOMES:
Psychological impact of the use of a social assistance robot on the child, his parents and his siblings | Visit 1 between Day 10 and Day 20 et visit 2 between Day 21 and Day 45
  psychological effects measured by semi-directive interviews of the parents and the brothers and sisters
Psychological effect of the use of a social assistance robot on the practice of nursing professionals in the service | Visit 2 between Day 21 and Day 45
  The effects will be explored through semi-structured interviews of nursing professionnals.

CONTACTS AND LOCATIONS:
Overall Officials: Rémi IZOULET, Principal Investigator — Toulouse Hospital

IPD SHARING:
Plan to Share IPD: No